CLINICAL TRIAL: NCT00106431
Title: A Single Agent Phase II Study of Depsipeptide (FK228) in the Treatment of Cutaneous T-cell Lymphoma
Brief Title: A Single Agent Phase II Study of Romidepsin (Depsipeptide, FK228) in the Treatment of Cutaneous T-cell Lymphoma (CTCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GPI-04-0001; NCT00337025 (obsolete NCT alias)
Record Dates: First submitted 2005-03-24; First posted 2005-03-25 (Estimated); Results first posted 2010-04-23 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Cutaneous T-cell Lymphoma
Keywords: romidepsin
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — romidepsin; Depsipeptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: romidepsin (depsipeptide, FK228) — Study patients received romidepsin at a dose of 14 mg/m^2 intravenously over 4 hours on Days 1, 8 and 15 of each 28-day cycle. The duration of study treatment was 6 cycles although patients who showed an objective response or stable disease could continue to receive therapy, at the discretion of the investigator, until disease progression or another withdrawal criterion was met.

SUMMARY:
GPI-04-0001 was a Phase II, non-randomized, open label, single arm study that was conducted at approximately 30 sites, primarily in the United States, Europe and Russia. It assessed the efficacy, safety, and tolerability of romidepsin as a treatment for cutaneous T-cell lymphoma (CTCL). Study patients (pts) received romidepsin in a dose of 14 mg/m^2 intravenously over 4 hours on Days 1, 8 and 15 of each 28-day cycle. The duration of study treatment was 6 cycles although pts who showed an objective response or stable disease could continue to receive therapy, at the discretion of the investigator, until disease progression or another withdrawal criterion was met.

DETAILED DESCRIPTION:
Responses were evaluated according to a composite assessment (Objective Primary Disease Response Evaluation Criteria [OPDREC]) that included cutaneous manifestations of disease, lymph node involvement, and circulating malignant T-cells (Sézary cells). Skin involvement was measured using a weighted body surface area skin assessment tool (WBSA/SWAT) or an erythroderma score, depending upon the pt's disease. Disease response was assessed by the Investigators and an Independent Response Review Committee (IRRC) with the IRRC assessment considered supportive of the Investigator's evaluations using the following criteria:

Complete Response (CR):

* Complete resolution of skin patches, skin plaques, and skin tumors, or erythroderma
* No evidence of abnormal lymph nodes
* Absence of circulating Sézary cells.
* No evidence of new tumors (cutaneous or non-cutaneous)
* Findings confirmed by skin biopsy

Clinical complete response (CCR):

- Same as CR but without skin biopsy

Partial Response (PR):

* ≥50% improvement in the summation of (change in Skin + change in Lymph Node + change in Peripheral Blood) with
* At least >30% improvement in Skin and
* No worsening in Lymph Node or Sézary cells.
* No evidence of new tumors (cutaneous/non-cutaneous)

Stable Disease (SD):

* Not enough improvement or worsening in the summation of (change in Skin + change in Lymph Node + change in Peripheral Blood to qualify as PR or PD
* No evidence of new tumors (cutaneous/non-cutaneous)

SD90:

- SD90 was defined as documented evidence of SD for at least 90 Days Duration

Progressive Disease (PD):

* Evidence of new tumor (cutaneous or non-cutaneous), OR
* >25% worsening in the summation of (change in Skin + change in Lymph Node + change in Peripheral Blood) with >15% worsening in change in Skin.

ELIGIBILITY:
Inclusion Criteria: Patients had to fulfill all of the following criteria to be eligible for study participation:

* Males or non-pregnant females aged 18 or over.
* Histologically confirmed diagnosis of CTCL, including mycosis fungoides and Sézary syndrome.
* Patients with CTCL stages II-A, II-B, III, and IV-A only.
* Patients with CTCL stage IB who had relapsed following previous therapy and where, in the investigator's opinion, the potential benefit of treatment with romidepsin outweighed the possible risks.
* Patients who had failed standardized skin-directed therapy and had had at least one course of systemic therapy, such as interferon, Ontak®, chemotherapy or Targretin®, etc., which they were deemed to have failed.
* Anticipated life expectancy greater than six months.
* Written informed consent to participate in the study.

Exclusion Criteria: Patients were ineligible for entry if any of the following criteria were met:

* ECOG Performance Status >1.
* Patients who had not received at least 1 course of prior systemic therapy for CTCL.
* Visceral involvement i.e. Stage 4B disease (lymphadenopathy was allowed).
* Patients with known cardiac abnormalities such as:

  * Congenital long QT syndrome
  * QTc (Corrected QT interval on ECG) interval >480 milliseconds
  * Any cardiac arrhythmia requiring anti-arrhythmic medication.
* Patients who had had a myocardial infarction within 12 months of study entry.
* Patients who had a history of coronary artery disease (CAD) e.g. angina Canadian class II to IV. In any patient in whom there was doubt, the patient should have had a stress imaging study and exercise electrocardiogram (ECG) and, if abnormal, angiography to define whether or not CAD was present.
* Patients with an ECG recorded at screening showing evidence of cardiac ischaemia (ST depression of >=2 mm). If in any doubt, the patient should have had a stress imaging study and exercise ECG and, if abnormal, angiography to define whether or not CAD is present.
* Patients with congestive heart failure that met New York Heart Association class II to IV definitions and/or ejection fraction <40% by multiple gated acquisition (MUGA) scan or <50% by echocardiogram and/or magnetic resonance imaging (MRI)
* Patients with a history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest, unless currently addressed with an automatic implantable cardioverter defibrillator (AICD).
* Patients with hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes (if in doubt, see ejection fraction criteria above).
* Patients with uncontrolled hypertension, i.e. >=160/95 mmHg.
* Concomitant use of any anti-cancer therapy.
* Concomitant use of warfarin (due to a drug interaction).
* Concomitant use of any investigational agent.
* Use of any investigational agent within 4 weeks of study entry.
* Concomitant use of drugs which may cause a prolongation of the QTc interval.
* Patients with a potassium level of <3.5 mmol/L and a magnesium level of <0.8 mmol/L.
* Clinically significant active infection.
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* Inadequate bone marrow or other organ function, as evidenced by:

  * unsupported haemoglobin <9.0 g/dL (transfusions and/or erythropoietin were permitted);
  * absolute neutrophil count (ANC) <=1.5 x 10^9/L;
  * platelet count <100 x 10^9/L;
  * total bilirubin >1.25 x upper limit of normal (ULN) for institution,
  * aspartate transaminase/glutamic oxaloacetic transaminase (AST/SGOT) and alanine transaminase/ glutamic pyruvic transaminase (ALT/SGPT) >2.0 x ULN, serum creatinine >2.0 x ULN for age and sex;
* Coexistent second malignancy or history of prior malignancy within previous 5 years (excluding basal or squamous cell carcinoma of the skin or cervical epithelial neoplasm [CIN1, carcinoma in situ] that had been treated curatively).
* Any significant medical or psychiatric condition that might have prevented the patient from complying with all study procedures.
* Patients who were pregnant or breast-feeding. All women of child bearing potential were to use an effective method of contraception (either an intrauterine device or a double barrier method using condoms or a diaphragm plus spermicide) during the study and for at least one month after receiving the last dose of romidepsin. Male patients were to use a barrier method of contraception (condoms) during the treatment period and for at least 1 month thereafter. Hormonal methods of contraception such as the contraceptive pill or patch (particularly those containing ethinyl estradiol) were to be avoided due to a potential drug interaction.
* Use of topical steroids in the previous 2 weeks or systemic steroids in the previous 4 weeks.
* Having previously given consent to participate in this study.
* Concomitant use of CYP3A4 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2008-06-01 (Actual); Study Completion 2008-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Nichols, Ph.D., Study Director — Gloucester Pharmaceuticals, Inc.
Locations (11):
- United States (6):
  - UCLA Jonsson Cancer Center, Los Angeles, California
  - Stanford Comprehensive Cancer Center, Stanford, California
  - Boston Medical Center, Boston, Massachusetts
  - University of Pennsylvania Abrahamson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Research Site, Multiple Locations, France
- Research Site, Multiple Locations, Germany
- Research Site, Multiple Locations, Poland
- Research Site, Multiple Locations, Russia
- Research Site, Multiple Locations, United Kingdom

REFERENCES:
- [Background] Duvic M, Bates SE, Piekarz R, Eisch R, Kim YH, Lerner A, Robak T, Samtsov A, Becker JC, McCulloch W, Waksman J, Whittaker S. Responses to romidepsin in patients with cutaneous T-cell lymphoma and prior treatment with systemic chemotherapy. Leuk Lymphoma. 2018 Apr;59(4):880-887. doi: 10.1080/10428194.2017.1361022. Epub 2017 Aug 30. PMID 28853310
- [Background] Foss F, Duvic M, Lerner A, Waksman J, Whittaker S. Clinical Efficacy of Romidepsin in Tumor Stage and Folliculotropic Mycosis Fungoides. Clin Lymphoma Myeloma Leuk. 2016 Nov;16(11):637-643. doi: 10.1016/j.clml.2016.08.009. Epub 2016 Aug 10. PMID 27637428
- [Background] Foss F, Coiffier B, Horwitz S, Pro B, Prince HM, Sokol L, Greenwood M, Lerner A, Caballero D, Baran E, Kim E, Nichols J, Balser B, Wolfson J, Whittaker S. Tolerability to romidepsin in patients with relapsed/refractory T-cell lymphoma. Biomark Res. 2014 Sep 8;2:16. doi: 10.1186/2050-7771-2-16. eCollection 2014. PMID 25279222
- [Background] Demierre M, et al. Pooled analyses of two international, multicenter clinical studies of romidepsin in 167 patients with cutaneous T-cell lymphoma (CTCL). Presented at 2009 ASCO Annual Meeting, May 29-June 2, 2009, Orlando, FL. Abstract No: 8546. J Clin Oncol 27:15s, 2009 (suppl)
- [Background] Cabell C, et al. Systematic Assessment of Potential Cardiac Effects of the Novel Histone Deacetylase (HDAC) Inhibitor Romidepsin. Presented at 2009 ASCO Annual Meeting, May 29-June 2, 2009, Orlando, FL. Abstract No: e19533. C J Clin Oncol 2009;27(suppl)
- [Background] Kim YH, et al. Clinically Significant Responses Achieved with Romidepsin in 37 Patient with Cutaneous T-Cell Lymphoma (CTCL) with Blood Involvement. Presented at American Society of Hematology 2009, New Orleans, LA. Abstract No. 2683.
- [Result] Whittaker SJ, Demierre MF, Kim EJ, Rook AH, Lerner A, Duvic M, Scarisbrick J, Reddy S, Robak T, Becker JC, Samtsov A, McCulloch W, Kim YH. Final results from a multicenter, international, pivotal study of romidepsin in refractory cutaneous T-cell lymphoma. J Clin Oncol. 2010 Oct 10;28(29):4485-91. doi: 10.1200/JCO.2010.28.9066. Epub 2010 Aug 9. PMID 20697094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between January 2005 and July 2007. Patients were enrolled at academic centers in the US and Europe that had experience in treating CTCL patients
Pre-assignment Details: Eligible patients were required to have failed at least 1 prior systemic therapy, e.g., interferon, chemotherapy, Ontak® (denileukin diftitox), or Targretin® (bexarotene).
Groups:
- Romidepsin: Regimen was 14 mg/m2 IV over a 4-hour period on Days 1, 8, and 15 of a 28-day cycle. The protocol included 6 cycles of treatment; responding patients and patients who achieved at least Stable Disease (SD) had the option of continuing treatment beyond 6 cycles at the discretion of the Investigator and based on local regulations.
Period: Overall Study
Arm/Group | Romidepsin
Started | 102
Completed | 37 (37 represents the number of patients who reached at least 6 months treatment)
Not Completed | 65

BASELINE CHARACTERISTICS:
Arm/Group | Romidepsin
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 79
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 62
Region of Enrollment [Number; unit: participants]
  France | 5
  United States | 20
  Poland | 24
  Russian Federation | 17
  Germany | 6
  United Kingdom | 20
  Georgia | 3
  Ukraine | 7
Eastern Cooperative Oncology Group (ECOG) Performance status [Number; unit: Participants]
  0, Fully active, able to carry on all pre-disease | 53
  1, Restricted in physically strenuous activity but | 49
  2, Ambulatory and capable of all selfcare but unab | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Patients (Pts) With Objective Disease Response
Description: The percent of pts with confirmed Objective Disease Response (confirmed best responses of complete response [CR], clinical complete response [CCR], or partial response [PR]). Responses were evaluated according to a composite assessment (Objective Primary Disease Response Evaluation Criteria - OPDREC).
Time Frame: 6 months
Population: Efficacy analysis based on interim analysis of data for as treated population
Measure: Number; unit: Percent of participants
Arm/Group | Romidepsin
Number analyzed (Participants) | 96
Percent of participants | 34

2. Secondary Outcome: Duration of Objective Disease Response
Description: Duration of Objective Response was defined as the number of months from the date of the first disease response (clinical complete response [CCR], or partial response [PR]) (later confirmed) until the date of progression and was determined using Kaplan-Meier product-limit estimates. In this analysis, pts who did not progress were censored as of their last evaluation with an OPDREC assessment.
Time Frame: Up to 10 months; median duration of follow up was 5.1 months
Population: Efficacy analysis based on interim analysis of data for as treated population
Measure: Median (Full Range); unit: Months
Arm/Group | Romidepsin
Number analyzed (Participants) | 96
Months | 14.91 [0.03 to 19.81]

3. Secondary Outcome: Time to Objective Disease Response
Description: Time to Objective Response was defined as the time in months from first dose date to the first date of objective disease response (later confirmed) and time to CCR was defined as the time in months from first dose date to the first date of CCR (later confirmed).
Time Frame: Up to 10 months
Population: Efficacy analysis based on interim analysis of data for as treated population
Measure: Median (Full Range); unit: Months
Arm/Group | Romidepsin
Number analyzed (Participants) | 96
Months | 1.87 [0.89 to 4.76]

4. Secondary Outcome: Time to Disease Progression
Description: Time To Progression was defined as the duration from the date of the first study drug dose to the date of progression (PD). In this analysis, pts who did not progress were censored at their last evaluation with an OPDREC assessment.
Time Frame: Up to 10 months; median duration of follow up was 6.1 months
Population: Efficacy analysis based on interim analysis of data for as treated population
Measure: Median (Full Range); unit: Months
Arm/Group | Romidepsin
Number analyzed (Participants) | 96
Months | 8.28 [0 to 21.65]

5. Secondary Outcome: Decrease in Pruritus Visual Analogue Scale (VAS) Score of ≥30 mm or a Score of 0 for at Least 2 Consecutive Cycles.
Description: Pruritus was reported monthly by pts using a 0 (no itching) to 100 (unbearable itching) mm visual analog scale (VAS). Pts were considered to have significant pruritus if the baseline VAS score was ≥ 30 mm. Clinically meaningful reduction in pruritus was defined as a decrease in VAS score of ≥ 30 mm or a score of 0 for at least 2 consecutive cycles.
Time Frame: Up to 10 months
Population: Patients meeting definition of moderate to severe pruritus on VAS (i.e., had a VAS of >=30 mm)
Measure: Number; unit: participants
Arm/Group | Romidepsin
Number analyzed (Participants) | 52
participants | 25

6. Secondary Outcome: Duration of Objective Disease Control (ODC)
Description: For pts with confirmed ODC (pts with CR, CCR, PR, SD90 [stable disease for 90 days]) based on OPDREC, duration of ODC was summarized with descriptive statistics, including number of censored observations, and 25th, 50th, 75th percentiles of distribution, based on Kaplan-Meier product limit estimates. For pts with confirmed progressive disease (PD), duration of ODC was calculated from first date of study drug to first date of diagnosis of confirmed PD. For pts without confirmed PD, duration of ODC was calculated from first date of study drug to date of the last visit with any OPDREC data.
Time Frame: Up to 10 months; median duration of follow up was 6.0 months
Population: Efficacy analysis based on interim analysis of data for as treated population
Measure: Median (Full Range); unit: Months
Arm/Group | Romidepsin
Number analyzed (Participants) | 96
Months | 17.67 [0.03 to 19.81]

7. Secondary Outcome: Percent of Pts With Objective Disease Control
Description: The percent of pts with confirmed ODC (CR, CCR, PR and SD90) based on OPDREC was summarized.
Time Frame: Up to 10 months
Population: Efficacy analysis based on interim analysis of data for as treated population
Measure: Number; unit: Percent of participants
Arm/Group | Romidepsin
Number analyzed (Participants) | 96
Percent of participants | 64

ADVERSE EVENTS:
Time Frame: Treatment emergent events were collected from first dose to last visit which occurred approximately 1 month after the last dose. Patients were to be treated for 6 cycles (approximately 6 months) or until progression.
Description: Patients could remain on treatment after 6 months if they experienced a response to treatment.
Arm/Group | Romidepsin
Serious Adverse Events (participants affected / at risk) | 23/102
Other Adverse Events (participants affected / at risk) | 99/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin (N=102)
Anaemia NOS (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Atrioventricular Block First Degree (Cardiac disorders) | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 1
Cardiac Failure NOS (Cardiac disorders) | 1
Cardiopulmonary Failure (Cardiac disorders) | 1
Cardiac Tamponade (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Colonic Perforation (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Rigors (General disorders) | 1
Pyrexia (General disorders) | 3
Disease Progression NOS (General disorders) | 2
Pain Exacerbated (General disorders) | 1
Oral Candidiasis (Infections and infestations) | 1
Oropharyngeal Candidiasis (Infections and infestations) | 1
Perineal Abscess (Infections and infestations) | 1
Sepsis NOS (Infections and infestations) | 3
Skin Bacterial Infection (Infections and infestations) | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1
Pharnygitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Electrocardiogram St Segment Depression (Investigations) | 1
Troponin I Increased (Investigations) | 1
Urine Output Decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1
Acidosis NOS (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neoplasm Progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Tumor Lysis Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Syncope (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Laryngeal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis Medicamentosa (Skin and subcutaneous tissue disorders) | 1
Haematoma NOS (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Hypotension NOS (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romidepsin (N=102)
Nausea (Gastrointestinal disorders) | 57
Vomiting NOS (Gastrointestinal disorders) | 35
Diarrhoea NOS (Gastrointestinal disorders) | 20
Constipation (Gastrointestinal disorders) | 12
Dry Mouth (Gastrointestinal disorders) | 7
Abdominal Pain NOS (Gastrointestinal disorders) | 6
Fatigue (General disorders) | 34
Pyrexia (General disorders) | 20
Asthenia (General disorders) | 14
Oedema Peripheral (General disorders) | 8
Lethargy (General disorders) | 6
Rigors (General disorders) | 5
Skin Infection (Infections and infestations) | 8
Upper Respiratory Tract Infection NOS (Infections and infestations) | 6
Blood Magnesium Decreased (Investigations) | 13
Haemoglobin Decreased (Investigations) | 7
Weight Decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 23
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Headache (Nervous system disorders) | 17
Dysgeusia (Nervous system disorders) | 15
Ageusia (Nervous system disorders) | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Anaemia NOS (Blood and lymphatic system disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 7
Hypotension NOS (Vascular disorders) | 7
Neoplasm Progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results at least 60 days prior to the date of submission for publication or public disclosure; sponsor will complete review within review period and will have authority to require institution/PI to delete confidential information other than the results.